CLINICAL TRIAL: NCT06974604
Title: Prevention of Datopotamab Deruxtecan (TROP-2 Directed ADC) Associated Stomatitis in Patients With HER2-negative Metastatic Breast Cancer or Non-small Cell Lung Cancer Using Dexamethasone Mouthwash: a Single-arm, Phase 2 Trial (TROPION- DM, 2023-ESR-000087)
Brief Title: Preventing Dato-DXd Associated Stomatitis With Dexamethasone Mouthwash, TROPION-DM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 431
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms; Lung Neoplasms
Keywords: Advanced/metastatic hormone-receptor positive [HR+], estrogen receptor and/or progesterone receptor positive; Advanced/metastatic triple negative breast cancer; Advanced/metastatic non-squamous, non-small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dexamethasone 10mL (Experimental): Prophylactic oral dexamethasone
  Interventions: Drug: Dexamethasone oral

INTERVENTIONS:
Drug: Dexamethasone oral — Dexamethasone 10 mL daily for days 1-5 for each of the ﬁrst 3 cycles of therapy Datopotamab Deruxtecan 6.0 mg/kg IV on day 1 every 21 days
  Other Names: Datopotamab Deruxtecan (Dato-DXd DS-1062a)

SUMMARY:
TROPION-DM/BrUOG-431 is a prospective, , phase 2 trial with two non-comparative cohorts analyzed jointly for primary endpoint in adult patients with either (Cohort 1:) advanced/metastatic hormone-receptor positive ([HR+], estrogen receptor and/or progesterone receptor positive) breast cancer (BC), or advanced/metastatic triple negative breast cancer (TNBC) or (Cohort 2:) advanced/metastatic non-squamous non-small cell lung cancer (NSCLC).

All patients will be treated with Datopotumab deruxtecan (Dato-DXd) at 6 mg/kg IV every 3 weeks until disease progression or unacceptable toxicity. Due to the risk of stomatitis, the investigational component of this trial will be to incorporate alcohol-free dexamethasone mouthwash, 10 mL 0.5 mg/5mL oral solution, days 1-5, swish and spit four times daily for the ﬁrst 3 cycles.

DETAILED DESCRIPTION:
See above summary

ELIGIBILITY:
Inclusion Criteria:

* Has advanced and/or metastatic cancer that meets one of the following criteria:

  1. Pathologically documented unresectable advanced non-squamous NSCLC not amenable to curative therapy that has progressed on at least one prior therapy.
  2. Pathologically documented triple negative breast cancer (estrogen receptor negative and progesterone receptor negative and HER2 negative) who have progressed on at least 1 prior line of therapy or in the opinion of the treating physician, not be a candidate for standard ﬁrst-line metastatic breast cancer therapy
  3. Pathologically documented hormone receptor positive breast cancer (estrogen receptor and/or progesterone receptor positive, HER2 negative) which has progressed on hormonal based therapy including CDK4/6 inhibitor and 1 prior line of chemotherapy and/or antibody drug conjugate therapy.
* Aged ≥18 years.
* Has an Eastern Cooperative Oncology Group performance status 0-2.
* Has a left ventricular ejection fraction (LVEF) 50% by either an echocardiogram (ECHO) or multiple gated acquisition scan (MUGA) within 28 days before enrollment.
* Measurable disease based on Response Evaluation Criteria in Solids Tumors (RECIST) version 1.1.
* Has adequate organ function that would make them an appropriate candidate for Datopotamab deruxtecan therapy as treatment of advanced metastatic cancer as assessed by the treating physician, which shall include results of complete blood count with diﬀerential, and comprehensive metabolic panel within 14 days before Cycle 1, Day 1, deﬁned as:

  1. Platelet count ≥100,000/mm3
  2. Hemoglobin ≥9.0 g/dL
  3. Absolute neutrophil count ≥1000/mm3
  4. Creatinine clearance ≥30 mL/min as calculated using the Cockcroft-Gault equation.
  5. Aspartate aminotransferase ≤3 ×ULN (if liver metastases are present, ≤5 × ULN)
  6. Alanine aminotransferase ≤3 × ULN (if liver metastases are present, ≤5 × ULN)
  7. Total bilirubin ≤1.5 × ULN if no liver metastases or liver < 3 if liver metastases are present.
* Has an adequate treatment washout period prior to Cycle 1, Day 1, deﬁned as appropriately recovering from:

  1. Major surgery: ≥2 weeks (or 2 weeks for low-invasive cases [eg, colostomy]).
  2. Radiation therapy (curative) and palliative radiation therapy to lung ﬁelds: ≥4 weeks; ≥2 weeks (palliative radiation therapy to other areas [ie, limited ﬁeld and 10 or fewer days or fractions] including whole brain radiotherapy).
  3. Hormonal therapy: ≥2 weeks
  4. Chemotherapy (including immunotherapy [non-antibody based therapy]), and retinoid therapy: ≥2 weeks or 5 times terminal elimination half-life (T½) of the chemotherapeutic agent (whichever is longer); ≥6 weeks for nitrosoureas or mitomycin C, ≥1 week for tyrosine kinase inhibitors (TKIs)
  5. Antibody-based anti-cancer therapy: ≥4 weeks
  6. Chloroquine/hydroxychloroquine: >14 days
* If of reproductive/child-bearing potential, agrees to use a highly eﬀective form of contraception or avoid intercourse throughout treatment and upon completion of the study for at least 7 months for females and 4 months for males after the last dose of study drug. Highly effective methods of birth control include: combined (estrogen and progesterone containing) hormonal contraception by oral or intravaginal route or dermal patches; progesterone-only hormonal contraception associated with inhibition of ovulation given by oral route or by injections or implants; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomized partner (with confirmation of surgical success); and complete heterosexual abstinence.
* Starting at the time of randomization/ﬁrst dose of study intervention male subjects/participants must not freeze or donate sperm at any time during this study and for at least 4 months after the last dose of Dato-DXd. Preservation of sperm should be considered prior to randomization/ﬁrst dose of study intervention.
* Starting at the time of randomization/ﬁrst dose of study intervention female subjects/participants must not breastfeed or donate, or retrieve for their own use, ova at any time during this study and for at least 7 months after the last dose of Dato-DXd. Preservation of ova should be considered prior to randomization/ﬁrst dose of study intervention.
* Is able to provide written informed consent and is willing and able to comply with the protocol. Subject must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible toxicities) and must sign and date the Institutional Review Board (IRB)/Independent ethics committee (IEC) approved informed consent form (ICF) (including Health Insurance Portability and Accountability Act authorization [HIPAA], if applicable) before performance of any study- speciﬁc procedures or examinations.
* Willingness to self-report level of oral pain using Visual Analog Scale (VAS) and the Normalcy Diet Scale (NDS) throughout each stomatitis event. (40, 41) At baseline, patient's self-reported oral pain level, using VAS, must be 0 (See Appendix B) and the normalcy diet scale score should ≥ 60 (See Appendix C).
* Willingness to record oral symptoms in Oral Diary (See Appendix D).
* Has a life expectancy of ≥3 months.

Exclusion Criteria:

* Active second malignancy which would alter interpretation of study results.
* Has a history of non-infectious ILD/pneumonitis including radiation pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has clinically signiﬁcant corneal disease
* Has a history of severe hypersensitivity reactions to either the drug or inactive ingredients (including but not limited to polysorbate 80) of Dato-DXd.
* Has a history of severe hypersensitivity reactions to other monoclonal antibodies.
* Has ongoing radiation-related toxicities
* Has an uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
* Has active human immunodeﬁciency virus (HIV) infection that is not well controlled.
* Has an active or uncontrolled hepatitis B and/or hepatitis C infection
* Is lactating or pregnant as conﬁrmed by pregnancy tests performed within 7 days before enrollment.
* Clinically severe pulmonary compromise resulting from autoimmune, connective tissue or inﬂammatory disorders with pulmonary involvement.
* Has uncontrolled or significant cardiac disease (including MI or unstable angina within the past 6 months, NYHA Class II-IV heart failure, uncontrolled hypertension, uncontrolled or significant arrhythmia).

Patients with the following may be enrolled based on the investigator's/treating physician's assessment (documentation must be submitted to BrUOG). -Mean resting corrected QTcF interval > 470 ms.

* History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
* Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Lower the incidence of all stomatitis | Approximately 9 weeks
  Lower the incidence of all stomatitis by 20%

SECONDARY OUTCOMES:
Clinical benefit | Approximately 9 weeks
  Clinical benefit rate

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Graff, MD, Principal Investigator — Rhode Island and the Miriam Hospitals (Brown University Health)
Locations (1):
- Rhode Island and the Miriam Hospitals (Brown University Health), Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No